CLINICAL TRIAL: NCT04645082
Title: Effect of Q-angle, Lateral Distal Tibial Angle and Proximal Muscle Torque on Ankle Injury
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Rabıa Tugba Kiliç, Doctor lecturer, Ankara Yildirim Beyazıt University
Other Study IDs: AYBU0507
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Ankle; Injury, Superficial, Multiple (With Foot)
Keywords: ankle injury, muscle strength, torque, knee, lower extremity
MeSH Terms: conditions — Wounds and Injuries; Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: x-ray examination — A total of 40 individuals who underwent an axial x-ray examination of the lower extremity following ankle sprain were included.

SUMMARY:
This study was undertaken to examine the effect of Q angle, lateral distal tibial angle (LDTA), and lower extremity isometric muscle torque on ankle sprain. Among 40 participants with ankle sprain, Q angle and LDTA measurements in both extremities were performed using X-ray images, while the muscle strength in gluteus maximus, gluteus medius, and quadriceps femoris were determined with hand held dynamometer, and the muscle torque was estimated by multiplying these values with the distance to the joint center. The obtained data were analyzed by separation analysis. No significant relationship was found between the Q angle and ankle sprain (p> 0.05). A strong positive correlation was found between LDTA and ankle sprain (p = 0.01). A strong negative correlation was found between quadriceps femoris muscle strength, gluteus medius muscle strength and gluteus maximus muscle strength with ankle sprain (p <0.001, p = 0.001, p <0.001, respectively). A strong negative relationship was found between quadriceps, gluteus medius and gluteus maximus muscle torques with ankle sprain (p <0.001, p = 0.011, p = 0.002, respectively). As suggested by the discrimination analysis, independent variables that contributed most to ankle injury included the gluteus maximus muscle torque (MAXIMUSTORQ) (.906), gluteus medius muscle torque (MEDIUSTORQ) (. 494), lateral distal tibial angle (.436) and quadriceps femoris muscle. torque (QUADRTORQ) (. 341), respectively. In conclusion, strengthening the quadriceps femoris, gluteus medius and gluteus maximus muscles may be suggested as an effective strategy to prevent ankle sprain. It may be helpful to pay attention to individuals with high LDTA to prevent ankle sprains.

DETAILED DESCRIPTION:
Ankle sprain is the most common type of ankle injury, comprising nearly 80% of all injuries affecting this area. Among these, 77% consists of sprains involving the lateral ankle (1). In sedentary individuals, the reported incidence is 5.2 to 6 per 1000 persons (2). Although the reported risk factors for ankle sprain include asymmetric tension in the flexor muscles of the ankle, increased body mass index (BMI), increased bodyweight, and younger age, definitive data is lacking (2).

The alignment of the pelvis, knee, and ankle has attracted significant research interest as a potential risk factor for lower extremity injury. Also, the quadriceps angle (Q angle) was reported to be an indicator for the biomechanical functions of the lower extremity, reflecting the effect of the quadriceps mechanisms on the knee, as well as providing information on patellar movements within the trochlear sulcus and on the functions of the thigh muscles (3). Q angle is measured as the narrow angle between the line that connects the anterior superior iliac spine (ASIS) to mid-patella and the line that connects the tibial tubercle with the center of patella (3, 4). Currently, no consensus exists regarding the normal value of the Q angle. While the American Orthopedics Society considers 10 degrees normal and 15 to 20 degrees as pathologic, the normal values reported by Schulthies et al. for males and females are 10 to 14 degrees, and 14.5 to 17 degrees, respectively (5). Several studies suggested that Q angle may actually represent an independent risk factor associated with increased risk of ankle sprain (4, 5). It has been proposed that individuals with knee valgus and a Q value exceeding 15 degrees have an increased risk of lower extremity injury. Also, a positive correlation between ankle sprain and Q angle was reported among recreational basketball players (3). On the other hand, no direct correlations were found between these two parameters in a study involving 45 professional athletes (4).

Another parameter that can be utilized to evaluate the alignment disorders of the lower extremity is the lateral distal tibial angle (LTDA). The average angle between the distal tibial joint orientation line and the anatomical and mechanical axis of the tibia is 89 degrees. This angle is referred to as LDTA (Figure 1). An angle of less than 86 degrees and more than 92 degrees indicate the presence of valgus and varus deformities, respectively (6). To the best of our knowledge, no previous studies have examined the association between LDTA and ankle sprain. It is plausible to assume that pathological LDTA, which is one of the alignment parameters of the lower extremity, may increase the predisposition to varus or valgus sprains. Therefore, our study was based on the hypothesis that LDTA may have an effect on the occurrence of ankle sprain, and thus it represents an intriguing research parameter. Also, when proximal muscle strength is assessed in people with chronic ankle imbalance, lack of muscle strength may be another potential risk factor for injury risk (9). This latter was particularly evident in studies that showed that the abductor muscle defects may lead to poor balance and neuromuscular adaptations in the ankle, therefore, contributing to increased inversion moments, increased activation, and earlier activation of the ankle evertors. When compared with athletes without injury, those with injury had weaker pelvic abduction and pelvic external rotation strength. In contrast, a prospective study by McHugh and colleagues concluded that the pelvic abductor, flexor or adductor strength had no role in predicting the future risk of ankle sprain (10).

Therefore, the published literature on the potential effects of Q angle on ankle sprain is controversial. On the other hand, literature data on the role of LDTA and proximal muscle strength on injury risk is also far from being clear. The primary objective of our study was to examine whether Q angle, LDTA, and knee and pelvic muscular torque were associated with ankle sprain. The secondary objective was to determine the parameter that had the most prominent impact on ankle injury risk.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with the lower extremity following ankle sprain were included.

Exclusion Criteria:

* Exclusion criteria were previous surgery of foot/knee and/or pelvis, age < 18 and > 65 years, presence of congenital/developmental lower extremity conditions, and other anomalies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with a lower limb ankle sprain
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Q angle | 5 months
  For Q angle measurements, the pivot of the goniometer was placed on the patella midpoint. One arm of the goniometer followed the longitudinal axis of the femur superiorly, while the other arm extended over the tibial tubercle on the tibia inferiorly It was performed on X-ray for Q angle measurement.
muscle strength | 5 months
  . The isometric muscular strength was measured with hand held dynamometer with the patient stabilized using external bents that precluded any movement of the muscle of concern for quadriceps femoris, gluteus medius and gluteus maximus muscles.
muscle torque | 5 months
  The distance between reference points were recorded in meters for muscle torque calculations. After completion of these measurements, the torque was estimated for the ankle with sprain and without sprain separately.
lateral distal tibial angle (LTDA) | 5 months
  LDTA was determined on the antero-posterior x-ray of the lower extremity by drawing a line on the anatomical axis of the tibia and another line for the distal tibial orientation, and LDTA was taken as the measure of the angle lateral to these two lines .

CONTACTS AND LOCATIONS:
Overall Officials: Mesut Uludag, Principal Investigator — Investigator; Ozge Vergili, Study Director — Director; Hayri Baran Yosmaoglu, Study Chair — Chair
Locations (1):
- Ankara Yildirim Beyazit University,Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There will be no IPD sharing plan.

REFERENCES:
- [Result] Guerra JP, Arnold MJ, Gajdosik RL. Q angle: effects of isometric quadriceps contraction and body position. J Orthop Sports Phys Ther. 1994 Apr;19(4):200-4. doi: 10.2519/jospt.1994.19.4.200. PMID 8173567